CLINICAL TRIAL: NCT00302835
Title: Case-Control Study on Analgesics and Nephropathy (SAN)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Other Study IDs: 2001_1
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Kidney Failure, Chronic
Keywords: Analgesics; Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

INTERVENTIONS:
Drug: non-phenacetin containing analgesics

SUMMARY:
The objective of the international, multicenter case-control study was to evaluate the association between end-stage renal disease (ESRD) and use of non-phenacetin-containing analgesics with particular emphasis on combined formulations.

DETAILED DESCRIPTION:
Background:

The association between intake of non-phenacetin-containing analgesics and the occurrence of chronic renal failure is still controversially discussed. A new epidemiologic study was planned and conducted in Germany and Austria.

Methods/design:

The objective of the international, multicenter case-control study was to evaluate the association between end-stage renal disease (ESRD) and use of non-phenacetin-containing analgesics with particular emphasis on combined formulations. A targeted sample of 1000 new (incident) dialysis patients, aged less than 50 years, was planned to recruit between January 1, 2001 and December 31, 2004. The age limit was chosen to avoid contamination of the study population with phenacetin-containing analgesics to the extent possible. Four control subjects per ESRD case, matched by age, sex, and region were selected from the population living in the region the case came from.

Lifetime exposure to analgesics and potential renal risk factors were recorded in a single face-to-face interview. A set of aids was introduced to reinforce the memory of study participants.

A standardized, pre-tested interview questionnaire (participants), a medical documentation sheet (physicians in dialysis centres), a logbook for all activities (dialysis centres) were used to collect the necessary data.

Quality management consisted of the standardized procedures, (re-) training and supervision of interviewers, regular checks of all incoming data for completeness and plausibility.

The study is scientifically independent and governed by a international Scientific Advisory Committee that bridged the gap between the sponsoring companies and the investigators. Also other advisory groups assisted the managing committee of the study. All relevant German and Austrian nephrological associations supported the study, and the study design was carefully reviewed and approved by the Kidney Foundation of Germany.

Discussion:

The study is expected to answer the main research question by end 2005. There is however a high potential for various biases that we tried to address with adequate measure. One limitation however cannot be overcome: The methodologically needed age-limitation of the study will make it not easy to generalize the results to age groups over 50 years. It might be suggested to repeat the study for persons over 50 years in 10 years when contamination with phenacetin use early in life is likely to be outgrown.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Patients under the age of 50 years with new (incident) chronic ESDR during the study period in a given dialysis center.
* Controls: Healthy persons from the same region the case came from and in the same 5-year age and gender group.

Exclusion Criteria:

* Patients with acute or remittent renal failure (e.g. after renal transplantation), out of age range, dead before the interview could be done, bad physical or mental condition

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4200
Dates: Start 2001-01; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Lothar AJ Heinemann, Professor, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Background] Heinemann LA, Garbe E, Lewis M, van der Woude F, Graf H. Case-control study on analgesics and nephropathy (SAN): protocol. BMC Nephrol. 2005 Aug 8;6:9. doi: 10.1186/1471-2369-6-9. PMID 16086834